CLINICAL TRIAL: NCT03874546
Title: Comparison Between the IMPACT's Score and the Clinician's Perception to Predict the Prognosis of Traumatic Brain Injury.
Brief Title: Comparison Between the IMPACT's Score and the Clinician's Perception to Predict the Prognosis of Severe and Moderate Traumatic Brain Injury
Acronym: PREDICT-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180477; 2018-A03135-50 (Other: ANSM)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury
Keywords: Severe and moderate traumatic brain injury; Prognosis; IMPACT score
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prognostic evaluation (Experimental): Questionnaire at Day1, Day7 and 6 months.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — * Two clinicians will complete a questionnaire that analyses their perception of the patient's prognosis at Day1 and Day7.
  * At 6 months, another clinician will establish the patient prognosis using Glasgow Outcome Scale and Glasgow outcome scale extended. This clinician must not know the patient's IMPACT score and prognosis established at Day 1 and Day 7. His evaluation will be compare to the patient's prognosis established previously (Day1 and Day7).
  Other Names: French language questionnaire for clinicians that analyses the clinician's perception of the patient's prognosis

SUMMARY:
Main objective : To compare the quality of the prognostic assessment, (adverse evolution at 6 months) of severe and moderate traumatic brain injury, performed by the clinician compared to the prognosis described by the IMPACT score.

The Pitié-Salpêtrière hospital is conducting a study evaluating the clinician's prognostic assessment of severe and moderate traumatic brain injury compared to the prognosis described by the IMPACT score. The investigators compare the quality of the clinician's prognostic assessment (adverse evolution at 6 months) of severe and moderate traumatic brain injury to the prognosis described by the IMPACT score.

DETAILED DESCRIPTION:
Design: Prospective, monocentric, pilot study. The study will be proposed to all patients admitted to the neurosurgical intensive care unit (ICU) at Pitié-Salpêtrière hospital, following a traumatic brain injury (TBI), over a period of 1 year. Around 100 patients will be included.

Day 1 : In the first 24 hours after traumatic brain injury, two clinicians will respond to the research questionnaire assessing their patient's prognosis, including confidence in their prediction and experience in neurological intensive care unit. The known prognostic variables as the IMPACT score in the first 24 hours will be collected.

Day 7 : The same clinicians will respond to the research questionnaire assessing their patient's prognosis, including confidence in their prediction and experience in neurological intensive care unit.

At 6 months : After 6 months, all patients or relatives will undergo a telephone interview (or if applicable during a follow-up visit in standard care) to assess the Glasgow Outcome Scale (GOS). This interview will be blinded to the clinician's prediction and the IMPACT score. For patients identified as GOS 3 or 4, a second GOS telephone interview will be carry out in the following days (<7 days), by a committee of adjudication composed of 2 examiners.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older,
* Hospitalized in the neurosurgical ICU department of the Pitié-Salpêtrière hospital following a head trauma,
* Presenting a Glasgow Coma Scale (GCS) ≤ 12 in the first 24 hours following the head trauma,
* Relatives informed of the research and not having objected to the patient's participation in the study.

Exclusion Criteria:

* Opposition of the patient,
* Patient under the protection of justice,
* Pregnant woman,
* Modified scale of Rankin> 1 before the traumatic brain injury.
* Patient unable to speak French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Compare the quality of the prognostic assessment of severe and moderate traumatic brain injury, performed by the clinician compared to the prognosis described by the IMPACT score. | At 6 month
  Comparison of the area under the ROC curve of the IMPACT model score for the prediction of the 6-month Glasgow Outcome Scale (GOS) ≤ 3 to the area under the ROC curve of the first day clinician's prediction.

SECONDARY OUTCOMES:
Differences in prognosis between clinicians based on their experience and specialty. | At 6 months
  Evaluation of the effect of the clinician's experience (number of years of neuro-ICU exercise) and specialty on the clinician's prognosis ROC curve.
To compare the quality of the prognosis of the clinicians between the 1st day (D1) and the 7th day (D7) post-traumatic. | At 6 months
  Comparison between the clinician's ROC curves at D1 (between the 6th and the 24th hour) and at D7 of the trauma for the prognosis of the patient.
Evaluate how the clinician's confidence in his prognosis is related to the quality of the prognosis. | At 6 months
  Evaluation of the effect of the clinician's confidence in his prognosis on the clinician's prognostic ROC curve.

CONTACTS AND LOCATIONS:
Overall Officials: Rémy BERNARD, MD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Réanimation neurochirurgicale, Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No